CLINICAL TRIAL: NCT01346449
Title: Making Calories Count: Information Format and Food Choice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 812950; P30AG034546 (NIH)
Record Dates: First submitted 2011-01-28; First posted 2011-05-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Obesity
Keywords: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Visual cue absent (Active Comparator)
  Interventions: Behavioral: Provide menu with no visual cue but with calorie information; Behavioral: Provide menu with no visual cue and no calorie information
- Calorie information present (Experimental)
  Interventions: Behavioral: Provide menu with visual cue and calorie information; Behavioral: Provide menu with no visual cue but with calorie information
- Calorie information absent (Active Comparator)
  Interventions: Behavioral: Provide menu with visual cue but no calorie information; Behavioral: Provide menu with no visual cue and no calorie information
- Visual cue present (Experimental)
  Interventions: Behavioral: Provide menu with visual cue and calorie information; Behavioral: Provide menu with visual cue but no calorie information

INTERVENTIONS:
Behavioral: Provide menu with visual cue and calorie information — Menu to be provided prior to placing the food order.
  Arms: Calorie information present; Visual cue present
Behavioral: Provide menu with visual cue but no calorie information — Menu to be provided prior to placing the food order.
  Arms: Calorie information absent; Visual cue present
Behavioral: Provide menu with no visual cue but with calorie information — Menu to be provided prior to placing the food order.
  Arms: Calorie information present; Visual cue absent
Behavioral: Provide menu with no visual cue and no calorie information — Menu to be provided prior to placing the food order.
  Arms: Calorie information absent; Visual cue absent

SUMMARY:
The purpose of the study is to better understand how individuals make decisions regarding the meals they order. Participants' ordering decisions at lunchtime at a chain restaurant will be recorded over several weeks to study ordering habits over time. Lunch menus will be provided by the study, and the menu format will vary the way in which information on caloric content is displayed.

The impact of different labeling formats on total calories in the chosen meal will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Customers of two chain restaurants

Exclusion Criteria:

* Unable to read a written menu

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Calories chosen | One time only or 6 months
  Total calories in food ordered for lunch

SECONDARY OUTCOMES:
Weight change | 6 months
  Half of the study participants will have the secondary outcome measure data collected and analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Julie Downs, PhD, Principal Investigator — Carnegie Mellon University
Locations (1):
- Carnegie Mellon University, Pittsburgh, Pennsylvania, United States